CLINICAL TRIAL: NCT05513365
Title: A Randomized Phase II Trial on the Addition of Dutasteride to Combined Androgen Blockade Therapy Versus Combined Androgen Blockade Therapy Alone in Patients With Recurrent and/or Metastatic Salivary Duct Carcinoma - DUCT Study
Brief Title: Phase II Dutasteride in Combination With CAB vs CAB in SDC
Acronym: DUCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MOHN22; 1140022110057 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-11

CONDITIONS: Salivary Duct Carcinoma
Keywords: Salivary duct carcinoma; Androgen deprivation therapy; Combined androgen blockade; Dutasteride; Goserelin; Bicalutamide; anti-androgens
MeSH Terms: interventions — Goserelin; bicalutamide; Dutasteride

STUDY DESIGN:
Intervention Model Description: Patients will be included into two cohorts based on their previous treatments, either ADT-naïve (cohort A) or ADT-resistant patients (cohort B). In cohort A, the randomization will result in the allocation of the control arm (goserelin and bicalutamide) and experimental arm (goserelin, bicalutamide, and dutasteride) in a 1:1 ratio. In cohort B, patients ADT-resistant will be enrolled receiving similar therapy to the experimental arm, i.e. goserelin, bicalutamide, and dutasteride.
  Cohort A is closed for inclusion as of April 18, 2024.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined androgen blockade (CAB) + dutasteride (Experimental): Patients from cohort B (ADT-resistant) will receive CAB+dutasteride.
  Interventions: Drug: Goserelin 10.8 mg; Drug: Bicalutamide 50 mg; Drug: Dutasteride 0.5 mg

INTERVENTIONS:
Drug: Goserelin 10.8 mg — Goserelin injection (10.8 mg) once per 3 months until progressive disease, intolerable toxicity, or investigator and/or patient decision to withdraw.
  Other Names: Zoladex
Drug: Bicalutamide 50 mg — Bicalutamide tablets (50 mg) once daily until progressive disease, intolerable toxicity, or investigator and/or patient decision to withdraw.
  Other Names: Casodex
Drug: Dutasteride 0.5 mg — Dutasteride capsules (0.5 mg) once daily until progressive disease, intolerable toxicity, or investigator and/or patient decision to withdraw.
  Other Names: Avodart

SUMMARY:
Phase 2 clinical trial on the addition of dutasteride to combined androgen blockade (CAB) therapy in recurrent and/or metastatic (R/M) salivary duct carcinoma (SDC) patients.

The study included two cohorts of patients: Cohort A, which comprises ADT-naïve patients, and Cohort B, which comprises ADT-resistant patients.

Cohort A is closed for inclusion as of April 18, 2024.

DETAILED DESCRIPTION:
A prospective, randomized controlled, single-institution, phase II clinical trial to assess the objective response rate (ORR), duration of response (DoR), progression free survival (PFS), overall survival (OS), toxicity, quality of life (QoL), and expression of molecular targets of patients with R/M SDC treated with either combined androgen blockade (CAB; goserelin + bicalutamide) or CAB + dutasteride, Participants in Cohort A will be randomized 1:1 at the study entry to receive CAB (goserelin 10.8 mg/3months + bicalutamide 50 mg/once daily) or CAB + dutasteride (0.5 mg/once daily). Participants will receive treatment until until progressive disease, intolerable toxicity, or investigator and/or patient decision to withdraw.

Cohort A is closed for inclusion as of April 18, 2024.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically/histologically proven diagnosis of (incurable) AR+ R/M salivary duct carcinoma
* AR positive diseases (strong expression in at least 1% of nuclei of neoplastic cells based on central IHC review)
* Measurable disease per RECIST version 1.1 at baseline. Appendix II.
* Age ≥ 18 years
* Written informed consent must be given according to national/local regulation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix III).
* Adequate bone marrow function:
* WBC ≥ 3.5/10^9 /L
* Absolute neutrophil count (ANC) ≥ 1.5x10^9/L
* Hemoglobin ≥ 6.20 mmol/L
* Platelet count ≥ 100x10^9/L
* Adequate liver function:
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN) OR ≤ 5.0 times ULN for patients with liver metastases
* Bilirubin ≤ 1.5 times ULN. For patients known with Gilbert's Syndrome ≤ 3.0 times ULN is permitted.
* Adequate renal function:
* Serum creatinine level ≤ 1.5 times ULN or calculated creatinine clearance ≥ 30 mL/min based on CKD-EPI-GFR
* Adequate cardiac function

Exclusion Criteria:

* Patients with history of allergic reactions attributed to compounds of similar chemical or biological composition to goserelin, bicalutamide or dutasteride
* Patients with peanut or soy allergy (dutasteride capsules contain lecithin which may contain soy oil)
* Patients who do not have adequate swallowing capacity
* Patients familiar with Long QT-syndrome (LQTS)
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measures
* Patients that are pregnant or lactating
* Patients with uncontrolled illness including:
* Cardiovascular disorders, including symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias
* Uncontrolled hypertension (defined as sustained systolic BP > 160 mm Hg, or diastolic BP > 100 mm Hg. Unless evidence of white-coat hypertension)
* Stroke (including TIA), myocardial infarction, or other ischemic event within 6 months before inclusion
* Serious active infections
* Patients undergoing concomitant treatments including:
* Concomitant (or within 4 weeks before inclusion) administration of any other experimental drug under investigation
* Concomitant (or within 6 months before inclusion) administration of any 5-alpha reductase inhibitor, i.e. dutasteride or finasteride
* Concurrent treatment with any other anti-cancer therapy within the last 4 weeks before inclusion
* Curative radiation therapy within the last 4 weeks before inclusion or palliative radiation therapy 1 week before start of study
* Any condition which, in the opinion of the investigator, would preclude participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Response will be measured according to RECIST version 1.1, the ORR is defined as the sum of the complete remissions plus partial responses. The best response will be used in each patient.
Duration of Response (DoR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Response will be measured according to RECIST version 1.1, the DoR is defined as the time from first tumor assessment at which the overall response was recorded as partial response (PR) or complete response (CR) that is subsequently confirmed until documented progressive disease (PD) or death form any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Response will be measured according to RECIST version 1.1, the PFS is defined as the time from study enrolment until date of first documented disease progression or death due to any cause, whichever occurs first.Every 12 weeks a CT/MRI scan will be made to asses the progression free survival until PD.
Clinical benefit rate (CBR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Response will be measured according to RECIST version 1.1, the CBR is defined as the confirmed CR or PR at any time or stable disease (SD) of at least 6 months. Every 12 weeks a CT/MRI scan will be made to asses the clinical benefit rate until PD.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The OS is defined as the time from study enrolment to the date of death to any cause.
Quality of Life (QoL) based on the EORTC QLQ-C30 questionnaire | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Quality of Life (QoL) based on the EORTC QLQ-C30 questionnaire. Participants are asked to fill in the questionnaires in week 0 (before start of treatment, baseline), every 12 weeks, and at PD.
Quality of Life (QoL) based on the EORTC QLQ-H&N43 questionnaire | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Quality of Life (QoL) based on the EORTC QLQ-H&N43 questionnaire. Participants are asked to fill in the questionnaires in week 0 (before start of treatment, baseline), every 12 weeks, and at PD.
Quality of Life (QoL) based on the EORTC QLQ-SHQ22 questionnaire | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Quality of Life (QoL) based on the EORTC QLQ-SHQ22 questionnaire. Participants are asked to fill in the questionnaires in week 0 (before start of treatment, baseline), every 12 weeks, and at PD.
Pain level assessed by the VAS (visual analog scale) questionnaire | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Scale range 0-10, in which a higher score represents more pain. Participants are asked to fill in the questionnaires in week 0 (before start of treatment, baseline), every 12 weeks, and at PD.
Adverse Events according to CTCAE v5.0 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Adverse events will be recorded using International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, the investigator will assess whether those events are drug related. Every OPD visit (every 3 months until PD)
Circulating tumor DNA (ctDNA) levels | through study completion, estimated after 3 years
  ctDNA levels will be assessed to evaluate whether treatment response and disease progression can be predicted. Baseline, 3 months, 6 months, and at PD.
mRNA expression levels of AR and AR splice variants | through study completion, estimated after 3 years
  mRNA expression of AR and AR splice variants on baseline and post-treatment tumor tissue samples to evaluate whether treatment response and disease progression can be predicted. Pre-treatment and post-treatment (i.e. PD)
mRNA expression levels of SRD5A1/SRD5A2 | through study completion, estimated after 3 years
  mRNA expression of SRD5A1/SRD5A2 on baseline and post-treatment tumor tissue samples to evaluate whether treatment response and disease progression can be predicted. Pre-treatment and post-treatment (i.e. PD)

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, prof. MD. PhD., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weijers JAM, Verhaegh GW, Lassche G, van Engen-van Grunsven ACH, Driessen CML, van Erp NP, Jonker MA, Schalken JA, van Herpen CML. A randomized phase II trial on the addition of dutasteride to combined androgen blockade therapy versus combined androgen blockade therapy alone in patients with advanced or metastatic salivary duct carcinoma - the DUCT study protocol. BMC Cancer. 2024 Sep 20;24(1):1174. doi: 10.1186/s12885-024-12889-0. PMID 39304797